CLINICAL TRIAL: NCT02863562
Title: Study of the Effect of Kinesio Taping and Proprioceptive Exercise on the Stability of Ankle in Amateur Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Inglés de la Torre, Principal investigator, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H1449680900364
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Injury of Musculoskeletal System

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): This group included 16 subjects. They received kinesio taping for both ankle joints and and performed proprioceptive exercises.
  Proprioceptive exercises were incorporated into their normal training routine (twice per week), and included 20 min of standardised proprioceptive exercises: single leg balancing on stable surfaces, on bosu/togu balls, and hopping activities, all repeated with eyes open/closed. Kinesio taping technique was used on both ankles on the first day of training with the aim of functional and mechanical correction, following the method described by Duenas et al. It was removed on the second day of training.
  Interventions: Other: Kinesio taping; Other: Proprioceptive exercises
- Group 2 (Experimental): This group received placebo kinesio taping for ankle joint (no tension) and performed proprioceptive exercises.
  Proprioceptive exercises were incorporated into their normal training routine (twice per week), and included 20 min of standardised proprioceptive exercises: single leg balancing on stable surfaces, on bosu/togu balls, and hopping activities, all repeated with eyes open/closed. Kinesio taping technique was used on both ankles on the first day of training in the same way as before but with no tension. It was removed on the second day of training.
  Interventions: Other: Proprioceptive exercises; Other: Placebo Kinesio taping
- Group 3 (Experimental): This group received kinesio taping for ankle joint. Kinesio taping technique was used on both ankles on the first day of training with the aim of functional and mechanical correction, following the method described by Duenas et al. It was removed on the second day of training.
  Interventions: Other: Kinesio taping

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping technique was used on both ankles on the first day of training with the aim of functional and mechanical correction, following the method described by Duenas et al. It was removed on the second day of training. This procedure was repeated each week for one month.
  Arms: Group 1; Group 3
Other: Proprioceptive exercises — Proprioceptive exercises were performed twice a week for one month. They were incorporated into their normal training routine (twice per week), and included 20 min of standardised proprioceptive exercises: single leg balancing on stable surfaces, on bosu/togu balls, and hopping activities, all repeated with eyes open/closed.
  Arms: Group 1; Group 2
Other: Placebo Kinesio taping
  Arms: Group 2

SUMMARY:
Soccer is a sport that attracts many participants and leads to a substantial number of injuries, especially of the ankle. Enhancement of functional joint stability by kinesio taping proprioceptive training may be important both in prevention and rehabilitation of ankle injuries. The main aim of this study was to determine the effect of kinesio taping and proprioceptive exercises on parameters related to ankle stability, such as the injury incidence, pain, static or dynamic stability and flexibility, in amateur soccer players training 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* To be older than 18 years old.
* To be soccer player for more than 5 years.

Exclusion Criteria:

* Serious illness.
* Recent ankle injury
* Vestibulocerebellar disorder
* Allergy to Kinesio taping
* Inability to complete all interventional sessions for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | 8 weeks
  Assessed by the Star Excursion Balance Test (SEBT). The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception. The goal of the SEBT is to maintain single leg stance on one leg while reaching as far as possible with the contralateral leg. Subjects are instructed to stand with both feet positioned inside the boundaries of the starting box. A trial initiates when the subject begins to reach in one of the four diagonal directions. In this study anterior, posteromedial and posterolateral directions will be evaluated. When reaching along the lines to the subject's right, the subject uses his right leg to reach while using his left leg as the support limb and vice versa. Subjects are not allowed to touch the ground with the reaching leg at any time during the reach. The maximal reach distance is the furthest point along the directional line.
Static balance | 8 weeks
  Assessed by the Unipedal Stance Test. Subjects are asked to close their eyes and to stand barefoot on the limb of their choice, with the other limb raised so that the raised foot is near but not touching the ankle of their stance limb. Prior to raising the limb, the subject is instructed to cross his arms over the chest. The investigator uses a stopwatch to measure the amount of time the subject is able to stand on one limb. Time commences when the subject raises the foot off the floor. Time ends when the subject either: (1) uses his arms (ie, uncrossed arms), (2) uses the raised foot (moves it toward or away from the standing limb or touches the floor), (3) moves the weight-bearing foot to maintain his balance (ie, rotates foot on the ground), (4) a maximum of 45 seconds has elapsed, or (5) opens eyes. The procedure is repeated 3 times and each time was recorded on the data collection sheet. The average of the 3 trials is recorded.
Flexibility | 8 weeks
  Assessed by the toe touch test. The subject stands on a box with his feet together and toes pointing forward. He is asked to bend from the hips forward and try to touch the ends of his fingers to the tips of your toes, without bending his knees. He should go as far as possible without pain, and try to keep his knees straight through the whole test. The distance to the basal line (top of the box) or over it is measured by a flexible tape.

SECONDARY OUTCOMES:
Pain | 8 weeks
  It was assessed by the FAAM questionaire (0= no pain; 10= great pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Marta Inglés, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dvorak J, Junge A. Football injuries and physical symptoms. A review of the literature. Am J Sports Med. 2000;28(5 Suppl):S3-9. doi: 10.1177/28.suppl_5.s-3. PMID 11032101
- [Background] Cruz-Diaz D, Lomas-Vega R, Osuna-Perez MC, Contreras FH, Martinez-Amat A. Effects of 6 Weeks of Balance Training on Chronic Ankle Instability in Athletes: A Randomized Controlled Trial. Int J Sports Med. 2015 Aug;36(9):754-60. doi: 10.1055/s-0034-1398645. Epub 2015 May 13. PMID 25969966
- [Background] Abian-Vicen J, Alegre LM, Fernandez-Rodriguez JM, Aguado X. Prophylactic ankle taping: elastic versus inelastic taping. Foot Ankle Int. 2009 Mar;30(3):218-25. doi: 10.3113/FAI.2009.0218. PMID 19321098
- [Background] Bicici S, Karatas N, Baltaci G. Effect of athletic taping and kinesiotaping(R) on measurements of functional performance in basketball players with chronic inversion ankle sprains. Int J Sports Phys Ther. 2012 Apr;7(2):154-66. PMID 22530190
- [Background] Han J, Anson J, Waddington G, Adams R, Liu Y. The Role of Ankle Proprioception for Balance Control in relation to Sports Performance and Injury. Biomed Res Int. 2015;2015:842804. doi: 10.1155/2015/842804. Epub 2015 Oct 25. PMID 26583139
- [Background] Akbari A, Sarmadi A, Zafardanesh P. The effect of ankle taping and balance exercises on postural stability indices in healthy women. J Phys Ther Sci. 2014 May;26(5):763-9. doi: 10.1589/jpts.26.763. Epub 2014 May 29. PMID 24926148
- [Background] Dueñas, L., Balasch, M., & Espí, G. (2010). Técnicas y nuevas aplicaciones del vendaje neuromuscular. Barcelona: Lettera Publicaciones.
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Background] Kinzey SJ, Armstrong CW. The reliability of the star-excursion test in assessing dynamic balance. J Orthop Sports Phys Ther. 1998 May;27(5):356-60. doi: 10.2519/jospt.1998.27.5.356. PMID 9580895
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175